CLINICAL TRIAL: NCT01594073
Title: Evaluation of Novel Biomarkers to Improve Risk Stratification and Patient Selection in ICD Therapy
Brief Title: Evaluation of Novel Biomarkers to Improve Risk Stratification and Patient Selection in Implantable Cardioverter-defibrillator (ICD) Therapy
Acronym: BIOMARKERICD
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Dr. David Duncker, Principal Investigator, Hannover Medical School
Other Study IDs: BIOMARKER-ICD
Record Dates: First submitted 2012-05-07; First posted 2012-05-08 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Ventricular Arrhythmias; Cardiac Death
Keywords: implantable defibrillator; ventricular arrhythmias; cardiac death
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma (EDTA, heparin), monocytes, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Implantable cardioverter-defibrillator (ICD) therapy reduces mortality in patients with chronic heart failure and reduced left ventricular ejection fraction (LVEF) <36%. Nevertheless, patient selection for ICD therapy based on LVEF and NYHA functional class alone seems to have a low specificity and sensitivity: In 100 patients treated, the SCD-HeFT study prevented 7 deaths in 5 years. Therefore 93 patients have a risk of adverse effects, such as operation risk, infection, pneumothorax, lead dislocation, and inadequate icd therapy. On the other hand, patients with advanced or end stage heart failure might rather die off progressive heart failure death and thus not benefit from ICD therapy.

It therefore seems appropriate and necessary to improve the individualized risk stratification in these patients. The aim of this study is to evaluate multiple cardiac biomarkers in a model predicting ventricular arrhythmias in patients on ICD therapy.

DETAILED DESCRIPTION:
Patients having or getting an ICD in the Dept. of Cardiovascular Medicine of the Hannover Medical School will be recruited in the next 2 years. Blood samples of all patients will be obtained at inclusion and at 6 months follow-up. Patients will be followed-up for 1-2 years after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient meeting the current indications for primary or secondary prophylactic ICD/CRT-D therapy
* age 18 years or older

Exclusion Criteria:

* Patient unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients reveicing or having received an implantable cardioverster-defibrillator in the Dept. of Cardiovascular Medicine of the Hanover Medical School.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-04; Primary Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
ICD therapy | 2 years
  ICD therapy (ATP/Shock) for ventricular fibrillation/ventricular tachycardia or inadequate therapy for supraventricular tachycardia/oversensing/lead dysfunction

SECONDARY OUTCOMES:
Quality of life | 2 years
  MLWHFQ, EQ5D
Depression scale | 2 years
  PHQ-9
6-Minute-walk-test | 6 months
  6-Minute-walk-test
all-cause mortality | 2 years
  All-cause mortality
Heart Failure Events | 2 years
  Changes in NYHA classification, Hospitalizations
Risc Scores for Heart Failure events/ICD therapy | 2 years
  Seattle Heart Failure Model, Lee-Score, PROFIT-Score

CONTACTS AND LOCATIONS:
Overall Officials: David Duncker, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany